CLINICAL TRIAL: NCT01529931
Title: Follow Up Study: The Effect Of Hair2Go Maintenance Treatments on Long Term Hair Removal
Brief Title: Long Term Efficiency of the Hair2Go Device
Acronym: OHR-8-FU-1Y
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OHR-8-FU-1Y; DC83411 (Other: Syneron Beauty)
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Hair Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (1):
- Maintenance (Experimental): This arm receives Hair2Go treatments once a month for 6 months
  Interventions: Device: Hair2Go

INTERVENTIONS:
Device: Hair2Go — Hair2Go treatment once a month for 6 months
  Other Names: Mē my elōs

SUMMARY:
The current study is a follow up study designed to gather information about the effect of the number of Hair2Go maintenance treatments on hair clearance 1 year after the last basic Hair2Go treatment. This study includes taking photos and documenting endpoints but does not include treatments.

DETAILED DESCRIPTION:
The Hair2Go device is intended for short-term and long-term removal of unwanted hair adjunctive to shaving. The device uses a technology called Elōs, which is a combination of electrical field at radio frequencies (RF) and intense optical energy, that are simultaneously applied to the tissue and were found to have synergistic effects. Thus, lower levels of both energies are used to facilitate the treatment for individuals of all skin types and hair colors.

This study is a multicenter study. Subjects that completed the basic treatments of previous Hair2Go studies (OHR-2, OHR-3, or OHR-5-Face) will be offered the option to enroll in this study that will not include treatments. The individual data collected in the OHR-2 (and its extensions, i.e. OHR2-P and OHR2-1Y), OHR-3, and OHR-5-Face studies will be used for the analysis together with data gathered in this study. Photographs of the previously treated areas will be taken 3, 6, 9, and 12 months after the last basic treatment if they were not already taken as part of the OHR-2, one of its extensions (i.e. OHR2-P and OHR2-1Y), or OHR-5-Face.

ELIGIBILITY:
Inclusion Criteria:

1. Completed the basic treatments of OHR-2, OHR-3, or OHR-5-Face studies.
2. Healthy males and females, between 18 and 65 years of age.
3. Willing to sign informed consent.
4. Willing to follow the protocol schedule.
5. Willingness to have photographs of the treated area taken that may be used for marketing and educational presentation and/or publications
6. Willingness to avoid shaving 1 week prior to the visits.

Exclusion Criteria:

1. Subject is taking medication that may have effect on hair growth (i.e. hormones, minoxidil)
2. Subject had electrolysis treatment within the last 6 months over the treatment area.
3. Subject had any type of professional intense pulsed light (IPL), laser or RF hair removal in the treatment site (with the exception of treatments within the OHR-2, OHR-2P, OHR2-1Y, OHR-3, or OHR-5-Face protocol).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Hair clearance at final follow up | 1 year after last basic treatment (termination)
  Hair clearance will be calculated at the final follow-up treatment from the hair counts conducted by independent blinded reviewer(s) based on photographs of treatment sites.

CONTACTS AND LOCATIONS:
Overall Officials: Jerome M Garden, MD, Principal Investigator — Northwestern Memorial Hospital; Vince Afsahi, MD, Principal Investigator — South Coast Dermatology Institute; Brian D Zelickson, MD, Principal Investigator — Abbot Northwestern Hospital Center for Cosmetic Care; Lilach Gavish, PhD — Hebrew University of Jerusalem
Locations (3):
- United States (3):
  - South Dermatology Institute, Tustin, California
  - Dr Jerome Garden, Chicago, Illinois
  - Zel Skin & Laser Specialists, Edina, Minnesota

IPD SHARING:
Plan to Share IPD: No
Only 5 subjects enrolled into this protocol. Data was combined with OHR2-1Y protocol and reported under that study.